CLINICAL TRIAL: NCT03614000
Title: Early Screening for Emotional, Behavioral and Autism Spectrum Disorders in Children With Functional Constipation.
Brief Title: Early Screening of Emotional, Behavioral and Autism Spectrum Disorders in Children With Functional Constipation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth Keuleneer, ASO Kinder- en Jeugdpsychiatrie, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: B.U.N. 143201733193
Record Dates: First submitted 2018-07-07; First posted 2018-08-03 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Functional Constipation; Emotional Problems; Behavioural Problems; Developmental Disorder; Autism Spectrum Disorder
Keywords: Childhood Constipation
MeSH Terms: conditions — Mental Disorders; Developmental Disabilities; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- positive screenings (Experimental)
  Interventions: Other: Screening Questionnaires

INTERVENTIONS:
Other: Screening Questionnaires — Measurement tools:
  * Social Responsiveness Scale (SRS-2) is a validated 65-item scale for the screening of ASD that requires parents to rate the child's behaviors in the previous 6 months. The questionnaire assesses interpersonal behavior, communication and repetitive/stereotypic behavior characteristics of ASD.
  * The Aseba Questionnaires are validated diagnostic tools that can be filled in by the parents, teachers or children to evaluate various behavioral and emotional problems. The CBCL assesses internalizing (i.e., anxious, depressive and over-controlled) and externalizing (i.e., aggressive, hyperactive, noncompliant and under-controlled) behaviors.
  * The VG&O The VG&O is a questionnaire developed in Dutch that gives a subscale of parental stress (OBVL), family functioning (VGFO), education habits (VSOG) and life events (VMG). The OBVL will be used

SUMMARY:
A significant group of children with functional constipation (FC) continues to have symptoms despite recommended standard therapy. Underlying psychiatric problems could explain therapy resistance. However, a work-up for psychiatric problems is only recommended after unsuccessful 6 months standard therapy. Earlier detection and check-up could lead to faster start-up of a more adequate therapy. Therefore, we investigate the prevalence of emotional, behavioural and social problems in the FC-population at the first contact with a paediatric gastroenterologist in a tertiary care hospital.

DETAILED DESCRIPTION:
The diagnosis of functional constipation (FC) in children leads to several diagnostic and therapeutic challenges. Most children respond well to standard recommended treatment, but there is a considerable group of patients that will continue to have symptoms. In this group, paediatricians sometimes presume the presence of an underlying psychopathology such as a developmental disorder, mood disorder, behavioural disorder. A longer treatment period has shown strong association with behavioural problems, suggestive for treatment resistant constipation.

It is known that functional defecation disorders (FDD) can be associated with behavioural and developmental disorders, such as Autism Spectrum Disorder (ASD) and Attention Deficit and Hyperactivity Disorder (ADHD), though these disorders are often initially unrecognized. Also, there are no clear guidelines reported regarding the timing when to search for underlying psychopathology in FC.

Research using Social Responsiveness Scale (SRS) and Social Communication Questionnaire-Lifetime (SCQ-L), screening tools for social difficulties, did not identify ASD diagnosis, in children with functional constipation. At the other hand, they found a total increase in emotional and behavioural problems in their research group. Prior studies found that 28 % of children with FDD referred to a tertiary centre scored positive on ASD screening questionnaires. A high prevalence of behavioural problems (37 %) in children with FC has been described as well.

According to the Guidelines for children with FC of the North American and European Societies of Paediatric Gastroenterology, Hepatology and Nutrition, the diagnosis of emotional, behavioural and/or developmental disorders (ASD or ADHD) will be considered after an unsuccessful six-month standard treatment.

We hypothesized that it could be useful to incorporate an earlier screening for emotional, behavioural and autism spectrum disorders into the diagnostic work-up of children with functional constipation referred to a tertiary care hospital. FC may have an important impact on the Quality of Life (QoL) in families of these children. Therefore we also measure parental stress and negative life-events from the child's perspective using the 'Opvoedingsbelasting Vragenlijst' (OBVL) for measurement of parental stress and the 'Vragenlijst Meegemaakte Gebeurtenissen' (VMG) for possible stressful life events from the child's perspective.

This study includes Dutch and French-speaking children, age 4-18 years, presenting for the first time at KidZ Health Castle (KHC) Brussels with suspicion of functional constipation complaints. Children could present ambulatory or could be hospitalized and were eligible regardless of previously diagnosed behavioural and developmental problems and regardless of any previous treatment for FDD. The diagnosis of FC was made based on the Rome IV criteria. Given that the 2 month interval listed in the Rome IV criteria for older children may unfairly delay treatment in some children with constipation, children who had difficulty with defecation for at least 2 weeks were also included 3. Children with an underlying organic cause that could have contributed to the development of constipation and children with functional non-retentive faecal incontinence (FNRFI) will be excluded.

The questionnaires will be given to the consenting parents and/or patients at the first visit and after 6 months conventional treatment along with an explanation of the research by the attending pediatrician, informed consent and a return envelope. Each questionnaire will be anonymized and provided with a code that will be linked to the name and number of the participant's file.

The group within the normal range at first visit for the two screening surveys: SRS-2 and CBC-L will serve as a control group.

Both groups will have to fill in the 2 questionnaires 6 months later, after initiation of adequate treatment. If the control results are still abnormal, participants will be directed to the department of Child and Adolescent Psychiatry for further treatment of their behavioral, emotional or developmental problems.

Participants will be seen every 2 - 3 months and outcome will be evaluated at 6 and 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting for the first time at the department of Pediatrics of the Universitair Kinderziekenhuis Brussel with complaints of constipation will be included regardless of previously diagnosed behavioral and developmental health problems and regardless of any previous treatment for functional defecation disorders.
* Developmental age 4-18 years
* Children and parents who express themselves fluently in Dutch or French
* Children who meet the Rome IV criteria for the diagnosis of functional constipation in children
* Children with developmental age of at least 4 years

At least two of the following present at least once per week for at least one month.

* Two or fewer defecations in the toilet per week
* At least one episode of fecal incontinence per week
* History of retentive posturing or excessive volitional stool retention
* History of painful or hard bowel movements
* Presence of a large fecal mass in the rectum
* History of large-diameter stools that may obstruct the toilet
* The symptoms cannot be fully explained by another medical condition.

Exclusion Criteria:

* Children with an underlying disease that could have contributed to the development of constipation: Celiac disease, Hypothyroidism, hypercalcemia, hypokalemia, Diabetes mellitus, Dietary protein allergy, Drugs, toxics, Vitamin D intoxication, Botulism, Cystic fibrosis, Hirschsprung Disease, Anal achalasia, Colonic inertia, Anatomic malformations, Pelvic mass (sacral teratoma), Spinal cord anomalies, trauma, tethered cord, Abnormal abdominal musculature (prune belly, gastroschisis, Downsyndrome), Pseudoobstruction (visceral neuropathies, myopathies, mesenchymopathies), Multiple endocrine neoplasia type 2B
* Children with functional non-retentive fecal incontinence (FNRFI).

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2021-08-12 (Estimated); Study Completion 2021-10-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of internalizing and externalizing behavioural problems as assessed by the Aseba questionnaires | 1 year
  The set of Aseba Questionnaires is a validated diagnostic tool that can be filled in by the parents, teachers or children to evaluate various behavioral and emotional problems. It assesses internalizing (i.e., anxious, depressive and over-controlled) and externalizing (i.e., aggressive, hyperactive, noncompliant and under-controlled) behaviors. It is the most widely used instrument for assessing child behavioral and emotional symptoms and can be converted into standardized scores (e.g., T scores Mean = 50, SD = 10) with higher scores indicating more emotional problems.
The prevalence of behavioural and social responsiveness problems as assessed by the Social Responsiveness Scale-2. | 1 year
  Social Responsiveness Scale (SRS-2) is a validated 65-item scale for the screening of ASD that requires parents to rate the child's behaviors in the previous 6 months. The questionnaire assesses interpersonal behavior, communication and repetitive/stereotypic behavior characteristics of ASD.

OTHER OUTCOMES:
The number of positive screens for parental stress as assessed by the OBVL questionnaires. | 1 year
  The OBVL is a part of the VG&O, a questionnaire developed in Dutch that gives information about parental stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Kinderziekenhuis Brussel, Jette, Brussels Capital, Belgium